CLINICAL TRIAL: NCT02379611
Title: Clinical Trial Comparing Neurologic Development of Temporal Voice Area in Cochlear Implanted Deaf Infant and in Normally Hearing Infant.
Brief Title: Study of Neurologic Development of Temporal Voice Area (TVA) in Deaf Infant
Acronym: Implaneuro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P130706; HAO13016 (Other: Assistance Publique)
Record Dates: First submitted 2014-12-19; First posted 2015-03-05 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Profound Congenital Deaf Children Implanted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- normally hearing children (Active Comparator)
  Interventions: Procedure: fNIRS (Functional Near Infrared Spectroscopy)
- Congenital profound deaf children (Experimental)
  Interventions: Procedure: fNIRS (Functional Near Infrared Spectroscopy)

INTERVENTIONS:
Procedure: fNIRS (Functional Near Infrared Spectroscopy) — fNIRS is a non-invasive imaging method involving the quantification of chromophore concentration resolved from the measurement of near infrared (NIR) light attenuation, temporal or phasic changes. NIR spectrum light takes advantage of the optical window in which skin, tissue, and bone are mostly transparent to NIR light in the spectrum of 700-900 nm, while hemoglobin (Hb) and deoxygenated-hemoglobin (deoxy-Hb) are stronger absorbers of light. Differences in the absorption spectra of deoxy-Hb and oxy-Hb allow the measurement of relative changes in hemoglobin concentration through the use of light attenuation at multiple wavelengths.

SUMMARY:
Hypothesis At 12 months of age, the neurologic development of TVA of a non cochlear implanted profound congenital deaf infant would be different to the development of a normally hearing infant.

At 24 months of age, the neurologic development of TVA of deaf infant implanted before the age of 18 months would be similar to the development of a normally hearing infant.

Main aim The main aim of the research is to study, by means of functional near infrared spectroscopy (fNIRS), the neurologic development of the TVA at 24 months of age (+/- 1 month) in a group (n=40) of normally hearing infant and in a group (n=40) of profound congenital deaf children implanted before the age of 18 months.

Main outcome Measure and localization of an increase of brain blood flow during an auditory stimulation "voice" type compared to a stimulation "non-voice" type. Comparison of the results between groups at 24 months of age +/- 1 month allows to analyse eventual differences.

Secondary aims and outcomes To study by means of functional near infrared spectroscopy the neurologic development of the temporal voice area at 12 months of age (+/- 1 month) in a group of normally hearing infant and in a group of profound congenital deaf infant wearing a standard hearing device between the age of 11 and 13 months and who will receive a cochlear implant between 12 and 18 months of age.

To study the association between fNIRS data and clinical data of the evaluation of comprehension of the spoken language at 24 months of age.

Methods Two groups of 40 infants matching in age will be constituted. Less than 13 months old children will be included during a medical consultation in the ENT department of Necker hospital after complete information of both parents. Written consent of both parents will be required. An audiophonological checking will be done.

Then a fNIRS examination will be programmed at the maternity of the Robert Debré hospital and done at the age of 12 months (+/- 1 month) and 24 months (+/-1 month). A fNIRS examination will be programmed at 36 months of age (+/- 1 month) for patinets included in the first year of the study.

This fNIRS examination measures the modifications in brain blood flow during the listening of human voice sound and environmental sound.

DETAILED DESCRIPTION:
One or two among a thousand new-born will require hearing device or cochlear implantation before the age of 4 years to correct a hearing loss. Without any appropriate hearing stimulation, some brain area, including temporal voice area (TVA), will remodel. But this remodeling process is a deleterious phenomenon in case of future cochlear implantation. Therefore it seems to be crucial to better understand the impact of hearing loss on neurologic development of TVA in infant.

Main aim and outcome:

Main aim of the research is to compare cortical activation in the TVA at 24 months of age (+/- 1 month), by means of the measure of hemoglobin and/or desoxyhemoglobin concentration in the TVA during listening of human voice sound compared to non-voice sound (environmental sounds) (fNIRS method):

* in normally hearing infants
* in profound congenital deaf infants who received a standard auditory device before the age of 10 months and who were implanted between 12 and 18 months of age.

Comparison of the results in these two groups at 24 months +/- 1 month will allow to evaluate the impact of hearing loss and of its rehabilitation by means of standard hearing device and then by cochlear implant on neurologic development of the TVA in infant.

Main outcome is the recording of a difference in the measure of hemoglobin and/or desoxyhemoglobin concentration during listening of human voice sounds compared to environmental sounds in the TVA, in both groups of infants at 24 months old (+/- 1 month). A difference in localization of activations in the "deaf" group would suggest a modification of the neuro-development of the TVA due to the hearing loss. On the contrary, a similar localization of activated areas would suggest a "picking up" of the neuro-development of TVA due to the correction of hearing loss by means of an auditory device.

Secondary aims and outcomes

Compare cortical activation in the TVA at 12 months of age (+/- 1 month) by means of the measure of hemoglobin and/or desoxyhemoglobin concentration in the TVA during listening of human voice sounds compared to environmental sounds:

* in normally hearing infants
* in profound congenital deaf infants who received a standard auditory device before the age of 10 months and who were implanted between 12 and 18 months of age.

Secondary outcome is the recording of a difference in the measure of hemoglobin and / or desoxyhemoglobin concentration in the TVA during listening of human voice sounds compared to environmental sounds in both groups of infants at 12 months of age (+/- 1 month).

Comparison of the results in these two groups at 12 months +/- 1 month will allow to evaluate the impact of hearing loss and of its rehabilitation by means of standard hearing device and then by cochlear implant on neurologic development of the TVA in infant.

Comparison of results obtained at 12 months (+/- 1 month) and 24 months (+/- 1 month) of age in both groups will allow the study of neurological development of TVA in normally hearing infants and in deaf infants wearing an auditory device for a period of one year.

Study association between development of oral communication, measured by means of questionnaire of evaluation of communication development and of comprehension of oral language in infant, and activation of TVA at 24 months of age by means of fNIRS.

ELIGIBILITY:
Inclusion criteria for deaf infants:

* child between 11 and 13 months at the time of the first fNIRS imaging testless
* Isolated congenital bilateral profound deafness
* Bilateral conventional hearing equipment between 2 and 10 months of life
* Rehabilitation project by cochlear implantation between 12 and 18 months accepted by parents
* French speaking parents
* Normal eardrums on otoscopy
* Signature of consent by both parents or by the sole parent with parental authority
* Beneficiary of a french social security (excluding AME)

Inclusion criteria for hearing infants:

* Any infant, followed in ORL consultation for any reason other than deafness, aged between 11 and 13 months at the time of the first fNIRS imaging examination.
* normal otoscopic examination
* Parents speaks French
* Signature of consent by both parents or by the sole parent with parental authority

Non inclusion criteria deaf infants:

* Stay in intensive care unit
* Premature birth
* Proven neuro-pediatric disorder
* Acquired deafness

Non inclusion criteria for hearing infants:

* Stay in intensive care unit
* Premature birth
* Proven neuro-pediatric disorder

Exclusion criteria for hearing infants:

- Acquired deafness during study

Max Age: 13 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Measure and localization of an increase of brain blood flow during an auditory stimulation "voice" type compared to a stimulation "non-voice" type at 24 months of age. | 24 months of age

SECONDARY OUTCOMES:
Measure and localization of an increase of brain blood flow during an auditory stimulation "voice" type compared to a stimulation "non-voice" type at 12 months of age. | 12 months of age
Brain blood flow by means of fNIRS (Functional Near infrared Spectroscopy) | 24 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Loundon, MD, Principal Investigator — Assistance Publique
Locations (1):
- Hôpital Necker Enfants malades Service d'ORL, Paris, France